CLINICAL TRIAL: NCT07276009
Title: The Effect of Multi-strain Probiotic Formulation on Gastrointestinal Symptoms, Quality of Life and Mental Health in Patients With Functional Dyspepsia: a Randomized Dietary Trial
Brief Title: Probiotics in Functional Dyspepsia
Acronym: ProPepsis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Biotic Sp. z o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MS-GIT-FD-A0004
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — Lacteol; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): L. rhamnosus LR110, B. lactis BI040, B. breve BB010, L. paracasei LPC100, L. acidophilus LA120, L. casei LR130, L. plantarum LP140, S. thermophilus ST250, B. longum BL020, B. bifidum BF030 5 billion CFU one time daily for 60 days
  Interventions: Other: Lactobacillus
- Placebo group (Placebo Comparator): Product with excepients without probiotic bacteria one time daily for 60 days
  Interventions: Other: Maltodextrin (Placebo)

INTERVENTIONS:
Other: Lactobacillus — 5 billion CFU of lactobacilus ans streptococci once daily for 60 days
  Arms: Probiotic group
Other: Maltodextrin (Placebo) — Placebo capsules will be given one a day for 60 days
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to learn whether a multi-strain probiotic can reduce digestive symptoms and improve quality of life in adults with functional dyspepsia. The main questions it aims to answer are:

* Does the probiotic reduce symptoms such as fullness after meals, bloating, stomach discomfort, and early satiation?
* Does the probiotic improve emotional well-being, including stress, anxiety, and mood? Researchers will compare the probiotic to a placebo (a look-alike capsule with no active ingredients) to see if the probiotic truly helps adults with functional dyspepsia.

Participants will:

* Take one capsule of the probiotic or placebo once daily before meals for 60 days
* Complete questionnaires about their digestive symptoms at the start, 1 month, and 2 months
* Complete surveys on stress, anxiety, depression, and quality of life at the start and 2 months
* Attend scheduled study visits for checkups and assessments

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Diagnosis of Functional Dyspepsia based on Rome IV criteria, with symptoms present for at least 3 months, and symptom onset at least 6 months before diagnosis, including:

   * Postprandial fullness
   * Early satiation
   * Epigastric pain or burning
   * (with no evidence of structural disease explaining symptoms)
3. Moderate to severe symptom severity at baseline, as defined by a validated scale (e.g., NDI or global symptom score)
4. Normal upper GI endoscopy within the last 12 months (or at screening), excluding structural disease (e.g., peptic ulcer, malignancy)
5. Negative for H. pylori (either previously treated successfully or tested negative within study screening)
6. Ability and willingness to provide informed consent and comply with study procedures
7. Stable medication use, if any, for at least 4 weeks before screening (e.g., PPIs, antidepressants, laxatives)

Exclusion Criteria:

1. Evidence of structural GI disease (e.g., peptic ulcer, gastric cancer, celiac disease) on recent or screening endoscopy
2. History of gastrointestinal surgery affecting stomach or small intestine (except appendectomy or cholecystectomy)
3. Positive test for H. pylori during screening (or untreated known infection)
4. Current or recent use (within 4 weeks) of antibiotics, pre-, pro- or postbiotics, unless part of study protocol
5. Use of medications affecting GI motility (e.g., prokinetics, opioids, anticholinergics) within 2-4 weeks before enrollment
6. Overlap with other functional GI disorders (except IBS) if they are the dominant complaint, unless your protocol allows overlap
7. Clinically significant psychiatric illness (e.g., major depression, schizophrenia) that may interfere with symptom reporting or adherence
8. Severe systemic or metabolic disease (e.g., uncontrolled diabetes, renal or hepatic failure)
9. Pregnancy or lactation, or intention to become pregnant during the study period
10. Participation in another clinical trial within the past 3 months
11. Known allergy or intolerance to study product components

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Gastrointestinal Symptom Rating Scale | 30 and 60 days

IPD SHARING:
Plan to Share IPD: Undecided